CLINICAL TRIAL: NCT02073890
Title: Incidence and Outcomes of Traumatic Subarachnoid Haemorrhage Patients: A Cross Sectional Study
Brief Title: Neurological Outcome in Patients of Traumatic Subarachnoid Haemorrhage
Status: Completed | Type: Observational
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: Center for Applied Research & Education (Unknown); SMS Medical College and Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CARE 1021/14
Record Dates: First submitted 2014-02-06; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Traumatic Subarachnoid Haemorrhage
Keywords: traumatic Subarachnoid Haemorrhage; Head Trauma; Computed Tomography
MeSH Terms: conditions — Subarachnoid Hemorrhage, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- traumatic subarachnoid haemorrhage

SUMMARY:
Traumatic brain injury is common cause of morbidity and mortality worldwide. Incidence and pattern of traumatic brain injury varies in developed and developing countries. Subarachnoid haemorrhage refers to blood in subarachnoid space that lies between arachnoid and piameninges, covering brain. It is often associated with concurrent intracranial injury component. Individuals at higher risk for tSAH are those who are at higher risk for blunt head trauma. This includes adolescents, low-income individuals, men, and individuals with a history of substance abuse. The investigators present study aims to investigate prognostic factors associated with the neurological outcome among patients of post traumatic SAH.

ELIGIBILITY:
Inclusion Criteria:

* All patients of traumatic subarachnoid haemorrhage

Exclusion Criteria:

* Metabolic disorder
* Altered coagulation profile
* Cardiac disease
* Co- morbid illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: traumatic subarachnoid haemorrhage
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Level of consciousness measured by Glasgow coma scale | Change from baseline to one month

SECONDARY OUTCOMES:
appearance of subarachnoid hemorrhage on CT measured by Fisher Grading | Change from baseline to one month

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Chair — Macmillan Research Group UK; Virendra D Sinha, M Ch, Study Director — SMS Medical College & Hospital, Jaipur; Manish Agrawal, M Ch, Principal Investigator — SMS Medical College & Hospital, Jaipur